CLINICAL TRIAL: NCT03621904
Title: PROMOTE Study: Prediction of Response Of HorMOnal Treatment in Advanced and Recurrent Endometrial Cancer
Acronym: PROMOTE
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Haukeland University Hospital (Other); Maastricht University Medical Center (Other); Brno University Hospital (Other); Holycross Cancer Center Kielce (Unknown); Medical University of Lublin (Other); Hospital del Mar (Other); Hospital Vall d'Hebron (Other); Royal Cornwall Hospitals Trust (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); The Netherlands Cancer Institute (Other); Canisius-Wilhelmina Hospital (Other); Catharina Ziekenhuis Eindhoven (Other); Erasmus Medical Center (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-3803
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-10

CONDITIONS: Endometrial Cancer Stage III; Endometrial Cancer Stage IV; Endometrial Cancer Recurrent
Keywords: Hormonal therapy; Endocrine therapy; Translational research; Tumor factors
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Antineoplastic Agents, Hormonal; Progesterone; Tamoxifen; Aromatase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Tumor samples originating from before start of hormonal therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- EC patients with HT: Patients with advanced stage or recurrent endometrial cancer treated with hormonal therapy
  Interventions: Drug: Hormonal Antineoplastics

INTERVENTIONS:
Drug: Hormonal Antineoplastics — Hormonal therapy used for treatment in endometrial cancer patients
  Other Names: Progesterone; Tamoxifen; Aromatase inhibitors

SUMMARY:
The PROMOTE study aims at optimising use of hormonal therapy in advanced stage and recurrent endometrial cancer analysing tumor tissue taken before start of hormonal therapy

DETAILED DESCRIPTION:
There is limited consensus about the position of hormonal treatment in advanced and metastatic endometrial carcinoma (EC). This is due to lack of good quality data on patient selection, and predictive biomarkers. Consequently, consideration of hormonal therapy is subjected to personal experience of the treating physician, rather than on refined clinical and up-to-date molecular criteria. Hormonal therapy has limited side-effects, and is better tolerated than systematic chemotherapy. Since EC patients are often elderly women with comorbidities, more effective and less aggressive treatment options are needed, underlining the urgency of an explorative study on this topic.

Endometrial cancer is the most common malignancy of the female genital tract in developed countries, with increasing incidence due to obesity and increased life expectancy. Most patients are diagnosed at an early stage, and have a favourable prognosis with surgery alone. Yet, 20% of the patients present with advanced or metastatic EC and have a poor outcome even with systemic treatment. Response rate of chemotherapy in advanced or metastatic EC is 30-60%, dependent of previous chemotherapy, with a progression free survival (PFS) of 3-14 months and 40% treatment related morbidity. In comparison, response to hormonal therapy is 20%-40%, with side effects in less than 5%. The overall PFS is 3 months, yet for those who respond the PFS can be up to several years.

To improve selective use of hormonal therapy in EC by evaluating applied hormonal therapy in advanced and metastatic EC and correlate response to molecular tumour analysis and translate this knowledge after validation into clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Advanced stage (FIGO stage III and IV) and recurrent endometrial cancer
* All histologic types of endometrial carcinoma
* Planned treatment with any type of hormonal therapy
* Biopsy taken within 120 days prior to start of hormonal therapy with no intercurrent therapy between biopsy and start of hormonal therapy.

Exclusion Criteria:

* Adjuvant hormonal therapy started following complete resection of endometrial carcinoma
* Synchronous use of hormonal therapy for other indications
* Endometrial sarcoma or endometrial stroma cell sarcoma

Ages: 18 Years to 110 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Endometrial cancer patients
Study Population: Patients with advanced stage and recurrent endometrial cancer treated with hormonal treatment, available biopsy prior to start of hormonal treatment and available follow-up
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Response rate | 2 years
  Complete or partial response according to RECIST criteria
Progression free survival | 2 years
  Interval from start of hormonal therapy to progressive disease or death
Clinical benefit rate | 2 years
  Complete or partial response or stable disease according to RECIST criteria

SECONDARY OUTCOMES:
Health-related quality of life | 6 months
  Health-related quality of life during hormonal therapy as tested with the validated EORTC-QLQ-C30 and EORTC-QLQ-EN24 quality-of-life scales at start of hormonal therapy and 6 months after start therapy

CONTACTS AND LOCATIONS:
Overall Officials: Hanny Pijnenborg, MD PhD, Principal Investigator — Radboud University Medical Center; Roy Lalisang, MD PhD prof, Principal Investigator — Maastricht University Medical Center; Andrea Romano, MD PhD, Principal Investigator — Maastricht University; Willem Jan Van Weelden, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
This is not yet established

REFERENCES:
- [Background] Amant F, Mirza MR, Koskas M, Creutzberg CL. Cancer of the corpus uteri. Int J Gynaecol Obstet. 2015 Oct;131 Suppl 2:S96-104. doi: 10.1016/j.ijgo.2015.06.005. No abstract available. PMID 26433681
- [Background] Moore TD, Phillips PH, Nerenstone SR, Cheson BD. Systemic treatment of advanced and recurrent endometrial carcinoma: current status and future directions. J Clin Oncol. 1991 Jun;9(6):1071-88. doi: 10.1200/JCO.1991.9.6.1071. PMID 2033421
- [Background] Fleming GF, Brunetto VL, Cella D, Look KY, Reid GC, Munkarah AR, Kline R, Burger RA, Goodman A, Burks RT. Phase III trial of doxorubicin plus cisplatin with or without paclitaxel plus filgrastim in advanced endometrial carcinoma: a Gynecologic Oncology Group Study. J Clin Oncol. 2004 Jun 1;22(11):2159-66. doi: 10.1200/JCO.2004.07.184. PMID 15169803
- [Background] Decruze SB, Green JA. Hormone therapy in advanced and recurrent endometrial cancer: a systematic review. Int J Gynecol Cancer. 2007 Sep-Oct;17(5):964-78. doi: 10.1111/j.1525-1438.2007.00897.x. Epub 2007 Apr 18. PMID 17442022
- [Background] Ethier JL, Desautels DN, Amir E, MacKay H. Is hormonal therapy effective in advanced endometrial cancer? A systematic review and meta-analysis. Gynecol Oncol. 2017 Oct;147(1):158-166. doi: 10.1016/j.ygyno.2017.07.002. Epub 2017 Jul 6. PMID 28689667
- [Background] Colombo N, Creutzberg C, Amant F, Bosse T, Gonzalez-Martin A, Ledermann J, Marth C, Nout R, Querleu D, Mirza MR, Sessa C; ESMO-ESGO-ESTRO Endometrial Consensus Conference Working Group. ESMO-ESGO-ESTRO Consensus Conference on Endometrial Cancer: Diagnosis, Treatment and Follow-up. Int J Gynecol Cancer. 2016 Jan;26(1):2-30. doi: 10.1097/IGC.0000000000000609. PMID 26645990
- [Background] Gibson WJ, Hoivik EA, Halle MK, Taylor-Weiner A, Cherniack AD, Berg A, Holst F, Zack TI, Werner HM, Staby KM, Rosenberg M, Stefansson IM, Kusonmano K, Chevalier A, Mauland KK, Trovik J, Krakstad C, Giannakis M, Hodis E, Woie K, Bjorge L, Vintermyr OK, Wala JA, Lawrence MS, Getz G, Carter SL, Beroukhim R, Salvesen HB. The genomic landscape and evolution of endometrial carcinoma progression and abdominopelvic metastasis. Nat Genet. 2016 Aug;48(8):848-55. doi: 10.1038/ng.3602. Epub 2016 Jun 27. PMID 27348297
- [Background] Vandenput I, Trovik J, Leunen K, Wik E, Stefansson I, Akslen L, Moerman P, Vergote I, Salvesen H, Amant F. Evolution in endometrial cancer: evidence from an immunohistochemical study. Int J Gynecol Cancer. 2011 Feb;21(2):316-22. doi: 10.1097/IGC.0b013e31820575f5. PMID 21734474
- [Background] Tangen IL, Onyango TB, Kopperud R, Berg A, Halle MK, Oyan AM, Werner HM, Trovik J, Kalland KH, Salvesen HB, Krakstad C. Androgen receptor as potential therapeutic target in metastatic endometrial cancer. Oncotarget. 2016 Aug 2;7(31):49289-49298. doi: 10.18632/oncotarget.10334. PMID 27384477
- [Background] Verhaegh W, van Ooijen H, Inda MA, Hatzis P, Versteeg R, Smid M, Martens J, Foekens J, van de Wiel P, Clevers H, van de Stolpe A. Selection of personalized patient therapy through the use of knowledge-based computational models that identify tumor-driving signal transduction pathways. Cancer Res. 2014 Jun 1;74(11):2936-45. doi: 10.1158/0008-5472.CAN-13-2515. Epub 2014 Apr 2. PMID 24695361
- [Background] Cornel KM, Kruitwagen RF, Delvoux B, Visconti L, Van de Vijver KK, Day JM, Van Gorp T, Hermans RJ, Dunselman GA, Romano A. Overexpression of 17beta-hydroxysteroid dehydrogenase type 1 increases the exposure of endometrial cancer to 17beta-estradiol. J Clin Endocrinol Metab. 2012 Apr;97(4):E591-601. doi: 10.1210/jc.2011-2994. Epub 2012 Feb 22. PMID 22362820
- [Background] Cornel KM, Krakstad C, Delvoux B, Xanthoulea S, Jori B, Bongers MY, Konings GF, Kooreman LF, Kruitwagen RF, Salvesen HB; ENITEC; Romano A. High mRNA levels of 17beta-hydroxysteroid dehydrogenase type 1 correlate with poor prognosis in endometrial cancer. Mol Cell Endocrinol. 2017 Feb 15;442:51-57. doi: 10.1016/j.mce.2016.11.030. Epub 2016 Dec 5. PMID 27923582